CLINICAL TRIAL: NCT03138252
Title: Randomized Controlled Trial: Cervical Ripening Balloon With and Without Oxytocin for Cervical Ripening in Multiparas
Brief Title: Study of the Effectiveness of Cervical Ripening Balloon With and Without Oxytocin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRB + Oxytocin
Record Dates: First submitted 2014-05-03; First posted 2017-05-03 (Actual); Results first posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Cervical Ripening; Induction of Labor; Multiparity
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cervical Ripening Balloon Alone (Active Comparator): Multiparous women will begin cervical ripening with a cervical ripening balloon alone. After the balloon is expelled or removed, induction of labor will proceed with pitocin per standard protocol at MacDonald Women's Hospital.
  Interventions: Drug: Oxytocin
- Cervical Ripening Balloon + Oxytocin (Active Comparator): Multiparous women will begin cervical ripening with a cervical ripening balloon and simultaneous oxytocin. After the balloon is expelled or removed, induction of labor will proceed with pitocin per standard protocol at MacDonald Women's Hospital.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin

SUMMARY:
Study Purpose: The purpose of this study is to determine the optimal method for induction of labor in multiparous women who present with an unfavorable cervix.

Hypothesis: Our hypothesis is that using oxytocin while the cervical ripening balloon is in place will result in more rapid labor courses, without increasing morbidity or increasing the need for operative delivery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Gestational age > 34 + 0/7 weeks
* Prior spontaneous vaginal delivery
* Clinical or U/S EFW of <4500 grams
* Singleton gestation
* Cervical dilation <2 cm

Exclusion Criteria:

* Any contraindication to cervical ripening balloon, pitocin, or vaginal delivery
* Placenta within 2 cm of cervical os
* Placental abruption, chorioamninoitis, or systemic infection prior to induction
* Rupture of membranes prior to induction ->1 prior C/S

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alison Bauer, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Cervical Ripening Balloon Alone: Multiparous women will begin cervical ripening with a cervical ripening balloon alone. After the balloon is expelled or removed, induction of labor will proceed with pitocin per standard protocol at MacDonald Women's Hospital.
  Oxytocin
- Cervical Ripening Balloon + Oxytocin: Multiparous women will begin cervical ripening with a cervical ripening balloon and simultaneous oxytocin. After the balloon is expelled or removed, induction of labor will proceed with pitocin per standard protocol at MacDonald Women's Hospital.
  Oxytocin
Period: Overall Study
Arm/Group | Cervical Ripening Balloon Alone | Cervical Ripening Balloon + Oxytocin
Started | 90 | 90
Completed | 90 | 90
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervical Ripening Balloon Alone | Cervical Ripening Balloon + Oxytocin | Total
Number analyzed (Participants) | 90 | 90 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 90 | 90 | 180
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 90 | 180
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 77 | 76 | 153
  White | 9 | 13 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 90 | 90 | 180

OUTCOME MEASURES:

1. Primary Outcome: Time From Cervical Ripening to Delivery
Description: Time from placement of cervical ripening balloon to delivery
Time Frame: Time to delivery
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cervical Ripening Balloon Alone | Cervical Ripening Balloon + Oxytocin
Number analyzed (Participants) | 90 | 90
hours | 16.88 [12.7 to 24.4] | 13.13 [10.8 to 17.7]

ADVERSE EVENTS:
Time Frame: 36 hours
Arm/Group | Cervical Ripening Balloon Alone | Cervical Ripening Balloon + Oxytocin
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90 | 2/90
Other Adverse Events (participants affected / at risk) | 0/90 | 0/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervical Ripening Balloon Alone (N=90) | Cervical Ripening Balloon + Oxytocin (N=90)
Peripartum Hysterectomy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 — Not study-related
Unanticipated neonatal intensive care unit admission (Pregnancy, puerperium and perinatal conditions) | 0 | 1 — Not study related

LIMITATIONS AND CAVEATS:
* Providers were not masked to the intervention group.
* We recruited 72%, but the inability to recruit all eligible patients is a potential source of selection bias.
* This study was not powered to assess adverse maternal/neonatal outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT03138252/Prot_SAP_000.pdf